CLINICAL TRIAL: NCT03972722
Title: An Open, Multi-center, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of Recombinant Fully Human Anti-PD-1 Monoclonal Antibody (GLS-010 Injection) in Patients With Recurrent or Metastatic Cervical Cancer
Brief Title: Study of GLS-010 Injection in Patients With Recurrent or Metastatic Cervical Cancer
Acronym: CC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH-S001-05
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLS-010 (Experimental): Full-human anti-pd-1 monoclonal antibodies
  Interventions: Drug: GLS-010

INTERVENTIONS:
Drug: GLS-010 — Patients will be given 240mg GLS-010 every treatment.
  Other Names: Full-human anti-pd-1 monoclonal antibodies

SUMMARY:
Patients with recurrent or metastatic cervical cancer，and will be treated with GLS-010.

DETAILED DESCRIPTION:
Open, uncontrolled, multi-center, phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the clinical trial; completely understanding and knowing about the study and signing the ICF; willingness and capability to comply with the requirements of the study.
2. Female aged from 18 to 75 years (margin included).
3. Cervical cancer patients with histologically confirmed PD-L1 positive (CPS ≥ 1).
4. Recurrent or metastatic cervical cancer patients who progress after receiving≥ 1 chemotherapy or are resistant to chemotherapy.
5. Based on RECIST 1.1, at least one measurable lesions, i.e. an extranodal lesion ≥10 mm in the longest diameter of cross-sectional areas or a lymph node lesion ≥ 15 mm in the shortest diameter of cross-sectional areas in CT or MRI test.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Life expectancy ≥ 12 weeks.
8. Organ and hematopoietic function as defined below:

   Hemoglobin (HGB) ≥ 90 g/L; White blood cell (WBC) ≥ 3 X 109/L; Absolute neutrophil count (ANC) ≥ 1.5 X 109/L; Platelets (PLT) ≥ 100 X 109/L; Total bilirubin≤ 1.5×upper limit of normal (ULN); AST and ALT ≤ 2.5×ULN or, for hepatic dysfunction due to liver metastases, ≤ 5×ULN; Serum creatinine (Cr) ≤ 1.5 X ULN or a creatinine clearance (CrCl) ≥ 50 mL/min; International normalized ratio (INR) or activated partial thromboplastin time (aPTT)≤1.5×ULN;
9. Female patients of childbearing potential should be willing to birth control after ICF signing, the course of the study, and 5 months after the last dose of study medication.
10. Patients must agree to provide either an archival tumor tissue sample or fresh biopsy sample for baseline biomarker tissue analyses, including staining for PD-L1. If archival tissue is not available and the patient does not have biopsy-accessible tumor lesions, the patient will be excluded.

Exclusion Criteria:

1. Prior therapy with an anti-PD1, anti-PDL1, anti-PDL2, anti-CD137 or anti-CTLA-4 agent (including Ipilimumab or any other drug specifically targeting T-cell co-stimulation or checkpoint pathways).
2. Prior anti-tumor therapy,(including chemotherapy, targeted small molecule therapy , radiotherapy, immunotherapy, mAb therapy) , or treatment with investigational products having not been launched onto the market in China in other clinical trials within 4 weeks prior to the first dose.
3. A past history of allergic reactions attributed to any macromolecular protein preparation/monoclonal antibody, or any other composition of the investigational product.
4. Pregnancy or lactation.
5. Patients with any autoimmune disease and received systemic therapy within 2 years (i.e. corticosteroids or immunosuppressive medications) [i.e.,but not limited to, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or caused by radiotherapy and chemotherapy can be included), patients with vitiligo or asthma CR in Childhood, not requiring any intervention in adulthood are permitted to enroll; patients with asthma requiring a bronchiectasis intervention are not permitted to enroll].
6. Subjects that requires systemic corticosteroids (dose equivalent to or above 10 mg prednisone daily) or other immunosuppressive medications within 14 days prior to enrollment or for the course of the study.
7. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Having received a live vaccine within 4 weeks prior to the first dose of investigational drug.
9. Having received a live anti-tumor vaccine, or anti-tumor treatment with immunostimulation.
10. Serious medical illness, such as severe infections, uncontrollable diabetes mellitus, cardiovascular diseases (i.e., grade 3 or 4 congestive heart failure (New York Heart Association (NYHA)), ≥ grade 2 heart block, myocardial infarction, uncontrolled arrhythmias, or unstable angina within 6 months prior to screening, and cerebral infarction within 3 months prior to screening) or lung diseases (i.e. interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm).
11. Patients with positive HBsAg and/or positive HBcAb with positive hepatitis B virus DNA> 103 copies/mL, or positive hepatitis C virus antibody; or positive syphilis.
12. A known history of human immunodeficiency virus (HIV) infection, or other acquired and congenital immune deficiency diseases.
13. A known history of active tuberculosis within 1 year prior to the first dose of investigational drug.
14. Presence of other malignant cancers within 5 years prior to enrollment. Patients with cured carcinoma in situ and cured skin basal cell carcinoma or cutaneous squamous cell carcinoma are eligible.
15. Having undergone allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
16. Having undergone major surgery (with the exception of baseline tumor biopsy), or serious trauma within 4 weeks prior to the first dose of therapy.
17. A history of alcoholism or drug abuse within 1 year.
18. A clear history of neurological or mental disorders, i.e. epilepsy, dementia, and poor compliance
19. Patients with other severe, acute or chronic disease that might increase risk of study drug use and participation, or laboratory abnormality that might confound the results of the trial.
20. Subjects not eligible for the study for other reasons, evaluated by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 89 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | within 27 Months after patient enrolled
  Based on an independent image assessment board

SECONDARY OUTCOMES:
PFS | within 27 Months after patient enrolled
  meaningful benefit in PFS based on RECIST 1.1
DCR | within 27 Months after patient enrolled
  meaningful benefit in DCR based on RECIST 1.1
DOR | within 27 Months after patient enrolled
  meaningful benefit in DOR based on RECIST 1.1
OS | within 3 years after patient enrolled.
  Overall survival
TTR | within 27 Months after patient enrolled
  meaningful benefit in TTR based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xia L, Wang J, Wang C, Zhang Q, Zhu J, Rao Q, Cheng H, Liu Z, Yin Y, Ai X, Gulina K, Zheng H, Luo X, Chang B, Li L, Liu H, Li Y, Lou G, Zhou Q, Zhu Y, Xiao Z, Tong J, Wang K, Chen J, Wang X, Song L, Wei Z, Ye Y, Zhu J, Wu X. Efficacy and safety of zimberelimab (GLS-010) monotherapy in patients with recurrent or metastatic cervical cancer: a multicenter, single-arm, phase II study. Int J Gynecol Cancer. 2023 Dec 4;33(12):1861-1868. doi: 10.1136/ijgc-2023-004705. PMID 37875323